CLINICAL TRIAL: NCT07394309
Title: A Phase I Pharmacokinetic Study of Hydronidone Capsules in Patients With Varying Degrees of Hepatic Impairment and Normal Hepatic Function.
Brief Title: Study of Hydroxynidone Capsules in Patients With Hepatic Impairment and Matched Healthy Controls
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KDN-F351-202507
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Liver Fibrosis
Keywords: Hydronidone; Liver Fibrosis; Patients with hepatic fibrosis due to chronic hepatitis B
MeSH Terms: conditions — Liver Cirrhosis | interventions — hydronidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group One A(mild hepatic impairment group) (Experimental): 10 participants with mild hepatic impairment (Child-Pugh A, score 5-6).
  Interventions: Drug: Hydronidone capsules
- Group Two B(moderate hepatic impairment group) (Experimental): 10 participants with moderate hepatic impairment (Child-Pugh Class B, score of 7-9).
  Interventions: Drug: Hydronidone capsules
- Group Three C（control group, normal hepatic function group） (Experimental): Matched 10 healthy participants with normal hepatic function will serve as the control group.
  Interventions: Drug: Hydronidone capsules

INTERVENTIONS:
Drug: Hydronidone capsules — A single oral dose of 90 mg of the investigational drug (3 Hydronidone capsules) under fasting conditions, administered with 240 mL of water.

SUMMARY:
This trial adopts a single-center, single-dose, open-label, non-randomized, parallel-controlled design. It will be conducted in participants with varying degrees of hepatic impairment, as well as in participants with normal hepatic function matched for sex, age, and BMI. The administration method is a single oral dose of 90 mg hydroxynidone capsules under fasting conditions.

Participants meeting the inclusion criteria with corresponding degrees of hepatic impairment and those with normal hepatic function will be enrolled. Each group will complete the study with 10 participants. Matched participants will be comparable in terms of sex (±1 participant per sex), mean age (±10 years), and mean BMI (±10%).

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be eligible for enrollment:
* Participants fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign a written informed consent form, and are able to complete the entire trial process as required by the protocol.
* Age between 18 and 75 years (inclusive), both males and females.
* At screening, male participants weigh ≥50 kg, female participants weigh ≥45 kg, and body mass index [BMI = weight (kg) / height² (m²)] is within the range of 18 to 32 kg/m² (inclusive).
* Participants and their partners agree to have no plans for conception or sperm/egg donation from the signing of the informed consent form until 6 months after the last dose of the investigational drug, and voluntarily agree to use effective contraceptive measures.
* Participants with hepatic impairment must additionally meet the following inclusion criteria:

Participants with hepatic impairment due to pre-existing primary liver disease, classified as Child-Pugh Class A (score of 5-6) or Class B (score of 7-9) at screening. They must not have received albumin infusion within 14 days prior to screening and must have a confirmed diagnosis of stable (≥1 month) hepatic impairment based on medical history, physical examination, laboratory tests, or imaging studies.

Participants have not taken any medication within 1 week prior to screening, or for those requiring long-term treatment for hepatic impairment and/or other comorbidities, their medication regimen must have been stable for at least 4 weeks (stability is judged by the investigator, excluding medications prohibited by the protocol).

Exclusion Criteria:

* Known history of allergy to any component of the investigational product, drugs of the same class (GLP-1 receptor agonists), or their excipients; or history of allergic constitution (multiple drug and food allergies); or history of allergic diseases (e.g., asthma, urticaria, eczematous dermatitis, etc.).
* Diagnosis of malignant tumor, or history of malignant tumor within 5 years prior to screening (except for: prior hepatocellular carcinoma surgery with stability ≥2 years; treated non-melanoma skin cancer with no signs of recurrence; and excised cervical intraepithelial neoplasia).
* Presence of severe infection, trauma, gastrointestinal surgery, or other major surgery within 4 weeks prior to screening.
* 12-lead electrocardiogram (ECG) abnormalities considered clinically significant by the investigator [e.g., tachycardia/bradycardia requiring medication, II-III degree atrioventricular block, prolonged QTcF interval (male QTcF >470 ms, female QTcF >480 ms, corrected using Fridericia's formula), or other abnormalities deemed clinically significant by the physician].
* Estimated glomerular filtration rate (eGFR) calculated using the Modification of Diet in Renal Disease (MDRD) formula <60 mL/min/1.73 m².
* Planned surgical procedure or hospitalization tendency during the trial period.
* Positive for HIV antibody (HIV-Ab) or Treponema pallidum (TP) antibody.
* Use of inducers or inhibitors of drug-metabolizing enzymes (CYP3A4 inducers and inhibitors, detailed list in Appendix 4: Common Drugs that are Inhibitors or Inducers of Drug-Metabolizing Enzymes) within 4 weeks prior to dosing.
* Use of drugs known to inhibit or induce SULT and UGT enzymes within 7 days prior to investigational drug administration, and inability to discontinue such use.
* Use of any medication (including herbal medicines, vitamins, health supplements) within 14 days (or 5 half-lives, whichever is longer) prior to dosing, except for stable medications in participants with hepatic impairment.
* Participation in another clinical trial and receipt of an investigational drug or medical device within 1 month prior to screening, with the last dose date of the previous clinical study as the reference point (if the previous investigational drug has a long half-life, at least 5 half-lives must elapse before dosing in this study).
* History of blood loss or blood donation ≥400 mL within 3 months prior to dosing, or plans to donate blood within 1 month after the end of this trial.
* History of smoking or smoking more than 5 cigarettes per day within 3 months prior to screening, or inability to abstain from any tobacco products during the study, or positive nicotine test at baseline.
* Regular alcohol consumption at present or within 1 month prior to screening, defined as females consuming more than 7 units of alcohol per week or males consuming more than 14 units of alcohol per week (1 unit = 285 mL of beer, or 25 mL of spirits with 40% alcohol, or 100 mL of wine); or positive alcohol breath test at baseline, or inability to abstain from alcohol during the trial.
* History of drug abuse, or use of soft drugs (e.g., marijuana) within 3 months prior to dosing, or use of hard drugs (e.g., cocaine, amphetamines, phencyclidine, etc.) within 1 year prior to dosing, or positive drug abuse screening at baseline.
* Consumption of food or beverages containing grapefruit juice/pomelo juice or methylxanthines (tea, coffee, cola, chocolate, energy drinks) within 48 hours prior to dosing, or consumption of any other substance that may affect drug absorption, distribution, metabolism, or excretion.
* Intolerance to venipuncture, history of needle phobia, or fainting at the sight of blood.
* Vaccination within 1 month prior to screening.
* Women who are pregnant or breastfeeding, or participants with a positive blood pregnancy test.
* Participants considered by the investigator to have poor compliance or other factors unsuitable for participation in this trial.
* Supplementary Exclusion Criteria for Participants with Hepatic Impairment (Exclusion if any one of the following criteria is met):

History of liver transplantation.

Drug-induced liver injury.

Acute liver injury due to any cause.

Cholestatic liver disease.

Liver failure with any of the following complications: uncontrolled infection; grade 3/4 hepatic encephalopathy.

Severe complications of cirrhosis with any of the following: active bleeding from esophageal or gastric varices; severe/advanced ascites or pleural effusion requiring paracentesis or drainage and albumin supplementation; hepatorenal syndrome; or any other condition deemed by the investigator as unsuitable for study participation.

Participants with poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg) or heart rate >120 bpm (allow two repeat measurements).

Any history of severe disease other than the primary liver disease itself, or any medical history or clinically significant abnormal laboratory findings considered by the investigator as likely to affect the trial results, including but not limited to history of circulatory, endocrine, neurological, digestive, urinary, hematological, immunological, psychiatric, or metabolic disorders.

Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >5 times the upper limit of normal (ULN) at screening.

Supplementary Exclusion Criteria for Participants with Normal Hepatic Function (Exclusion if any one of the following criteria is met):

Positive for anti-hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg).

History of primary disease of vital organs, including but not limited to neurological/psychiatric, cardiovascular, gastrointestinal, respiratory, urinary, endocrine, hematological, or immune system diseases, deemed by the investigator as unsuitable for trial participation.

History of hepatic impairment, or any screening examination results (including physical examination, vital signs, complete blood count, urinalysis, blood biochemistry, coagulation function, 12-lead ECG, chest X-ray posteroanterior view, abdominal ultrasound, etc.) considered by the investigator as clinically significant abnormalities.

Age not within the range of the mean age of participants with mild/moderate hepatic impairment ±10 years, and/or BMI not within the range of the mean BMI of participants with mild/moderate hepatic impairment ±10%.

-Supplementary Exclusion Criteria for Participants with Normal Hepatic Function (Exclusion if any one of the following criteria is met):

Positive for anti-hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg).

History of primary disease of vital organs, including but not limited to neurological/psychiatric, cardiovascular, gastrointestinal, respiratory, urinary, endocrine, hematological, or immune system diseases, deemed by the investigator as unsuitable for trial participation.

History of hepatic impairment, or any screening examination results (including physical examination, vital signs, complete blood count, urinalysis, blood biochemistry, coagulation function, 12-lead ECG, chest X-ray posteroanterior view, abdominal ultrasound, etc.) considered by the investigator as clinically significant abnormalities.

Age not within the range of the mean age of participants with mild/moderate hepatic impairment ±10 years, and/or BMI not within the range of the mean BMI of participants with mild/moderate hepatic impairment ±10%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter of Hydronidone: Cmax | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone: AUC0-t | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone:AUC0-∞ | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone:Tmax | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone:t1/2 | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone:λz | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone:CL/F | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone:MRT | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone:Vz/F | Within 48 hours of administration
Pharmacokinetic Parameter of Hydronidone:Ratio of free drugsRatio of free drugs | Within 48 hours of administration
Difference in the main parameters AUC₀-t between patients with hepatic impairment and participants with normal hepatic function. | Within 48 hours of administration
Difference in the main parameters AUC₀-∞ between patients with hepatic impairment and participants with normal hepatic function. | Within 48 hours of administration
Difference in the main parameters Cmax between patients with hepatic impairment and participants with normal hepatic function. | Within 48 hours of administration

SECONDARY OUTCOMES:
Plasma Pharmacokinetic Parameters of Metabolites M3 and M4: Cmax (Metabolic Ratio). | Within 48 hours after administration
Plasma Pharmacokinetic Parameters of Metabolites M3 and M4: AUC₀-t, (Metabolic Ratio). | Within 48 hours after administration
Plasma Pharmacokinetic Parameters of Metabolites M3 and M4: MR (Metabolic Ratio). | Within 48 hours after administration
Plasma Pharmacokinetic Parameters of Metabolites M3 and M4: AUC₀-∞, (Metabolic Ratio). | Within 48 hours after administration
Plasma Pharmacokinetic Parameters of Metabolites M3 andM4:Tmax(Metabolic Ratio). | Within 48 hours after administration
Plasma Pharmacokinetic Parameters of Metabolites M3 and M4: t₁/₂(Metabolic Ratio). | Within 48 hours after administration

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui, China